CLINICAL TRIAL: NCT06107959
Title: Changes in Resting Metabolic Rate Following Orthopedic Surgery
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Lisa Vopat, MD, Principal Investigator, University of Kansas Medical Center
Other Study IDs: STUDY00150689
Record Dates: First submitted 2023-10-12; First posted 2023-10-30 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Metabolism; Disorder, Postprocedural; Resting Metabolic Rate; Post Operative Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine Specific Gravity, hydration assessment in order to complete the body composition test.
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Male: 50 male subjects undergoing orthopedic surgery.
  Interventions: Other: Pre-surgical nutrition, hydration, RMR, and body composition assessments; Other: Post-surgical nutrition, hydration, RMR and body composition assessments
- Female: 50 female subjects undergoing orthopedic surgery
  Interventions: Other: Pre-surgical nutrition, hydration, RMR, and body composition assessments; Other: Post-surgical nutrition, hydration, RMR and body composition assessments

INTERVENTIONS:
Other: Pre-surgical nutrition, hydration, RMR, and body composition assessments — Urine sample, InBody device platform, Metabolic cart with hood to collect RMR.
Other: Post-surgical nutrition, hydration, RMR and body composition assessments — Same as pre-surgical tests at 1 week, 3 weeks, 6 weeks, and 12 weeks follow up time points.

SUMMARY:
This project is intended to determine the magnitude and duration of RMR changes in patients receiving orthopedic surgery. The result will help to guide postoperative nutrition recommendations in patients receiving orthopedic surgery.

DETAILED DESCRIPTION:
Surgery produces a catabolic response in the body that shifts metabolism from glucose to fat and protein. Despite no studies examining ACLR, studies of other orthopedic surgeries demonstrate increased postoperative energy expenditure, as well as a shift to beta-oxidation. Additionally, in most patients, these changes reverted to baseline within six weeks, although a subset of patients did not return to baseline until beyond 12 weeks.

This project will improve our understanding of magnitude and duration of RMR changes following orthopedic surgery, and the subsequent perioperative dietary suggestions that should be made to improve patient outcomes. Currently, postoperative dietary suggestions are not surgery nor patient specific. Determining how orthopedic surgery effects RMR will help to personalize perioperative treatment, rehabilitation, and recovery.

Better understanding the change in RMR following orthopedic surgery and implementing more accurate dietary modifications will help to ensure positive outcomes and control of infection following orthopedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Any individual over 15 undergoing an orthopedic surgery.

Exclusion Criteria:

* Pregnant female
* < 15 years old

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be over the age of 15 years old undergoing elective orthopedic surgery at KU Medical Center.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To determine the magnitude of the change in RMR of patients receiving orthopedic surgery. | 12 weeks
  RMR = (9.99 X actual weight*)+ (6.25 X height*) - (4.92 X age) - 161*use weight in kilograms (kilogram), height in centimeters (cm).
To observe the amount of time it takes the RMR to return to baseline. | 12 weeks
  calculation in number of weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braga M, Baccari P, Scaccabarozzi S, Fiacco E, Radaelli G, Gallus G, DiPalo S, DiCarlo V, Cristallo M. Prognostic role of preoperative nutritional and immunological assessment in the surgical patient. JPEN J Parenter Enteral Nutr. 1988 Mar-Apr;12(2):138-42. doi: 10.1177/0148607188012002138. PMID 3283387
- [Background] Hu SS, Fontaine F, Kelly B, Bradford DS. Nutritional depletion in staged spinal reconstructive surgery. The effect of total parenteral nutrition. Spine (Phila Pa 1976). 1998 Jun 15;23(12):1401-5. doi: 10.1097/00007632-199806150-00019. PMID 9654632
- [Background] Lenke LG, Bridwell KH, Blanke K, Baldus C. Prospective analysis of nutritional status normalization after spinal reconstructive surgery. Spine (Phila Pa 1976). 1995 Jun 15;20(12):1359-67. PMID 7676333
- [Background] Ljungqvist O, Soop M, Hedstrom M. Why metabolism matters in elective orthopedic surgery: a review. Acta Orthop. 2007 Oct;78(5):610-5. doi: 10.1080/17453670710014293. No abstract available. PMID 17966019
- [Background] Malone DL, Genuit T, Tracy JK, Gannon C, Napolitano LM. Surgical site infections: reanalysis of risk factors. J Surg Res. 2002 Mar;103(1):89-95. doi: 10.1006/jsre.2001.6343. PMID 11855922
- [Background] McMulkin ML, Ferguson RL. Resting energy expenditure and respiratory quotient in adolescents following spinal fusion surgery. Spine (Phila Pa 1976). 2004 Aug 15;29(16):1831-5. doi: 10.1097/01.brs.0000134564.24874.10. PMID 15303030